CLINICAL TRIAL: NCT06496087
Title: Evaluation of DEPREXIL Treatment in Patients With Clinical Depression Through Psychological and Neuroendocrine Assessment
Brief Title: Evaluation of DEPREXIL in Patients With Clinical Depression Through Psychological and Neuroendocrine Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEPREXIL_DEPRESSION_CO_2022
Record Dates: First submitted 2024-06-05; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Depression; Post-COVID-19 Syndrome; Depression Mild; Depression Moderate
Keywords: Depression; Antioxidant; Supportive Care; Post-COVID-19 Syndrome; Ginkgo Biloba
MeSH Terms: conditions — Depression; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deprexil Group (Experimental): The trial group will be administered 1 capsule of DEPREXIL orally every 8 hours for 6 months of treatment.
  Interventions: Dietary Supplement: DEPREXIL

INTERVENTIONS:
Dietary Supplement: DEPREXIL — The trial group will be administered 1 capsule of DEPREXIL orally every 8 hours for 6 months of treatment.

SUMMARY:
Clinical depression is a mood disorder that affects people of all ages with symptoms such as sadness, anger or frustration, appetite changes, difficulty concentrating and suicidal thoughts. Psychological and pharmacological treatments are available to treat it, such as cognitive behavioral therapy and antidepressants. Deprexil® from Catalysis is a food supplement that regulates neuronal metabolism and calcium homeostasis, which may help in cases of mild to moderate depression. It is proposed to conduct a study in patients with primary, secondary or post-COVID-19 depression to evaluate the effects of this supplement on psychological and neuroendocrine changes.

DETAILED DESCRIPTION:
Clinical depression is a mood disorder where feelings of sadness, anger or frustration interfere with daily life for a prolonged period of time. It can affect people of all ages, presenting symptoms such as irritable or low mood, difficulty falling asleep or oversleeping, change in appetite, fatigue, feelings of worthlessness, hatred and guilt, difficulty concentrating, and suicidal thoughts; however, in children these symptoms can vary, especially focusing on behavior, sleep, and school performance. Various treatments are available, ranging from psychological treatments, such as cognitive behavioral therapy or psychotherapy, to antidepressant medications, such as selective serotonin reuptake inhibitors, depending on the severity of the depression.

Deprexil® by Catalysis is a food supplement to treat mild and moderate depressive states. The molecular action process to which its active ingredients are subjected regulates neuronal metabolism as well as calcium homeostasis. A large number of diseases with an imbalance in calcium homeostasis have depressive effects on the Central Nervous System (CNS) and peripheral nervous system (PNS), and therefore, it is capable of regulating neuronal metabolism by stabilizing the neuronal membrane and favoring its oxygenation. Therefore, to evaluate the effects of Deprexil®, the investigators propose to conduct a study in patients diagnosed with primary depression or secondary to concomitant pathologies or post-COVID-19, treated with this dietary supplement, assessing psychological and neuroendocrine changes.

Each patient will undergo an initial evaluation by means of a psychological consultation, which will be carried out again 3 and 6 months after the beginning of the treatment. Likewise, the levels of hormones and neuropeptides such as GABA, Dopamine, Serotonin, Noradrenalin, Melatonin, Glutamate, Cortisol and dehydroepiandrosterone will be analyzed at the beginning and at the end of the treatment, which will consist in the intake of Deprexil® of Catalysis, in doses of three capsules daily during 6 months. Based on this, the correspondence with neuroendocrine alterations found in the patients will be evaluated according to the results of the psychological evaluation, seeking to evaluate the changes on the patient's symptomatology at clinical and paraclinical level, giving as results the analysis on the changes caused at neuroendocrine level secondary to COVID-19, to a concomitant pathology or to a primary depressive pathology.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical depression diagnosed primary or secondary to concomitant illness or post COVID-19.

Exclusion Criteria:

* Patients with psychological disorders in addition to depression, such as anxiety, attention deficit, hyperactivity disorder, post-traumatic stress disorder other than that caused by COVID-19, bipolar disorder or other mental disorders secondary to depression.
* Patients with severe depression requiring antidepressant medication.
* Patients who ingest psychoactive substances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
To evaluate the psychological state of depressive patients treated with Deprexil® by patient questionnaire test | 6 months
  To evaluate the psychological state of depressive patients treated with Deprexil® by Zung test of patients with a depressive state assessment tool using a Google Forms questionnaire, automatically tabulating the answers for analysis. Evaluation before, after 3 months and 6 months of treatment with Deprexil.
  Each item of the Zung scale can provide a score between 1 and 4; the range of values is therefore 20-80 points.
  1. Less than 28 points = No depression.
  2. between 28 and 41 points = Mild depression.
  3. between 42 and 53 points = Moderate depression.
  4. 53 or more points = Severe depression.
To evaluate the psychological state of depressive patients treated with Deprexil® by hormonal levels | 6 months
  To evaluate the psychological state of depressive patients treated with Deprexil®. To evaluate the concentration of hormones by means of NeuroSpot Kit in depressive patients before and after 6 months of treatment with Deprexil®. Kit will measure Serotonin, Creatinine, Dopamine, Noradrenaline, Adrenaline.
  Urine sample:
  • Second morning urine: The next urine over the course of the morning after getting up and after the first morning urine (Going to the toilet during the night does not count in this content)
  Saliva samples:
  * 1st Sample 0,5 hours after getting up
  * 2nd Sample at 12:00 noon
  * 3rd Sample at 8:00 PM
  Serotonin(55-129 ug/g creatinine) Dopamine (125-250 ug/g creatinine) Noradrenaline (25-55 ug/g creatinine) Adrenaline (3.0-7.0 ug/g creatinine)
To evaluate the psychological state of depressive patients treated with Deprexil® by hormonal levels | 6 months
  To evaluate the psychological state of depressive patients treated with Deprexil®. To evaluate the concentration of hormones by means of NeuroSpot Kit in depressive patients before and after 6 months of treatment with Deprexil®. Kit will measure Cortisol (morning, noon, evening).
  Urine sample:
  • Second morning urine: The next urine over the course of the morning after getting up and after the first morning urine (Going to the toilet during the night does not count in this content)
  Saliva samples:
  * 1st Sample 0,5 hours after getting up
  * 2nd Sample at 12:00 noon
  * 3rd Sample at 8:00 PM
  Cortisol (4.0-12; 1.5-5 ng/ml)
To evaluate the psychological state of depressive patients treated with Deprexil® by hormonal levels | 6 months
  To evaluate the psychological state of depressive patients treated with Deprexil®. To evaluate the concentration of hormones by means of NeuroSpot Kit in depressive patients before and after 6 months of treatment with Deprexil®. Kit will measure DHEA (morning, evening).
  Urine sample:
  • Second morning urine: The next urine over the course of the morning after getting up and after the first morning urine (Going to the toilet during the night does not count in this content)
  Saliva samples:
  * 1st Sample 0,5 hours after getting up
  * 2nd Sample at 12:00 noon
  * 3rd Sample at 8:00 PM
  DHEA (104-578; 45-251 pg/ml)
To evaluate the psychological state of depressive patients treated with Deprexil® by neuropeptides | 6 months
  To evaluate the psychological state of depressive patients treated with Deprexil®. To evaluate the concentration of neuropeptides by means of NeuroSpot Kit in depressive patients before and after 6 months of treatment with Deprexil®. Kit will measure GABA and Glutamate levels.
  Urine sample:
  • Second morning urine: The next urine over the course of the morning after getting up and after the first morning urine (Going to the toilet during the night does not count in this content).
  Saliva samples:
  * 1st Sample 0,5 hours after getting up
  * 2nd Sample at 12:00 noon
  * 3rd Sample at 8:00 PM
  GABA (2.25-12.8 umol/ g creatinine) Glutamate (8.0-30 umol/ g creatinine)

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación CR INVESTIGATION INSTITUTE, Bogotá, Bogotá DC, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Mazza MG, De Lorenzo R, Conte C, Poletti S, Vai B, Bollettini I, Melloni EMT, Furlan R, Ciceri F, Rovere-Querini P; COVID-19 BioB Outpatient Clinic Study group; Benedetti F. Anxiety and depression in COVID-19 survivors: Role of inflammatory and clinical predictors. Brain Behav Immun. 2020 Oct;89:594-600. doi: 10.1016/j.bbi.2020.07.037. Epub 2020 Jul 30. PMID 32738287
- [Background] Perez-Cano HJ, Moreno-Murguia MB, Morales-Lopez O, Crow-Buchanan O, English JA, Lozano-Alcazar J, Somilleda-Ventura SA. Anxiety, depression, and stress in response to the coronavirus disease-19 pandemic. Cir Cir. 2020;88(5):562-568. doi: 10.24875/CIRU.20000561. PMID 33064695
- [Background] Li Y, Scherer N, Felix L, Kuper H. Prevalence of depression, anxiety and post-traumatic stress disorder in health care workers during the COVID-19 pandemic: A systematic review and meta-analysis. PLoS One. 2021 Mar 10;16(3):e0246454. doi: 10.1371/journal.pone.0246454. eCollection 2021. PMID 33690641
- [Background] Mazza MG, Palladini M, Poletti S, Benedetti F. Post-COVID-19 Depressive Symptoms: Epidemiology, Pathophysiology, and Pharmacological Treatment. CNS Drugs. 2022 Jul;36(7):681-702. doi: 10.1007/s40263-022-00931-3. Epub 2022 Jun 21. PMID 35727534